CLINICAL TRIAL: NCT03495401
Title: Effect of Double Fortification (Iron and Zinc) in Synbiotic Milk to Under 5 Years Stunted Children Growth : the Efforts to Achieve Target 2 SDGs Utilizing Local Natural Resources
Brief Title: Effect of Double Fortification (Iron and Zinc) in Synbiotic Milk to Under 5 Years Stunted Children Growth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, DR.Siti Helmyati, DCN, M.Kes, DR., Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KE/FK/0640/EC/2017
Record Dates: First submitted 2018-03-04; First posted 2018-04-12 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Stunting
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Intervention Model Description: Intervention group given fortified synbiotic milk, control group given non-fortified synbiotic milk
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fortified synbiotic milk (Experimental): 100 ml fortified (7,47 mg ferrous sulphate and 4,33 mg zinc acetate) synbiotic milk containing 7 billion CFU Lactobacillus plantarum Dad13 in combination with 4 g prebiotic fructooligosaccharides
  Interventions: Dietary Supplement: fortified synbiotic milk
- non-fortified synbiotic milk (Placebo Comparator): 100 ml non-fortified synbiotic milk containing 7 billion CFU Lactobacillus plantarum Dad13 in combination with 4 g prebiotic fructooligosaccharides
  Interventions: Dietary Supplement: non-fortified synbiotic milk

INTERVENTIONS:
Dietary Supplement: fortified synbiotic milk — 100 ml fortified (7,47 mg ferrous sulphate and 4,33 mg zinc acetate) synbiotic milk containing 7 billion CFU Lactobacillus plantarum Dad13 in combination with 4 g prebiotic fructooligosaccharides
  Other Names: susu synbio (synbio milk) fortified
  Arms: fortified synbiotic milk
Dietary Supplement: non-fortified synbiotic milk — 100 ml non-fortified synbiotic milk containing 7 billion CFU Lactobacillus plantarum Dad13 in combination with 4 g prebiotic fructooligosaccharides
  Other Names: susu synbio (synbio milk) non-fortified
  Arms: non-fortified synbiotic milk

SUMMARY:
The purpose of this study is to investigate the effects of double fortification (iron and zinc) in synbiotic milk (L.plantarum Dad13 and fructooligosaccharides) on under 5 years stunted children growth, gut microbiota composition, blood zinc and hemoglobin level, and cognitive level.

DETAILED DESCRIPTION:
This is a parallel, quadruple-blind, randomized controlled trial to determine the effects of double fortification (iron and zinc) in synbiotic milk (containing 7 billion CFU L.plantarum Dad13 and 4 g fructooligosaccharides) on the gut microbiota composition, body height and weight, blood zinc and hemoglobin level, and cognitive level in under 5 years stunted children subjects. The duration of the study is 4 months, including a 2-week pre test and informed consent before randomization of subjects into treatment or control group, a 12-week intervention period, and a 2-week post test after the end of intervention. During the intervention period, subjects will be instructed to take 100 ml of fortified synbiotic milk or non-fortified synbiotic milk per day. They will also be asked to document consumed milk, any unusual symptoms or side effects of treatment. Diet will be monitored via 24-h dietary recalls and SQ-FFQ before and after treatment respectively. Changes in the gut microbiota composition will be determined by measuring bacterial population levels (Bifidobacteria, Lactobacillus, Enterobacteria, Prevotella, and Bacteroides) in stool sampled collected at baseline and 12 weeks by qPCR. Metabolic markers (calprotectin, hemoglobin, and zinc level) will be measured at baseline and 12-weeks in serum and plasma using biochemical and immuno-assay. Changes in the cognitive level, height for age Z-score collected at baseline and 12 weeks using Bayley Scales of Infant Development, 2nd Edition .

ELIGIBILITY:
Inclusion Criteria:

* age between 2 year to 5 years
* height per age z-score under -2 (stunting)
* parents sign inform consent form

Exclusion Criteria:

* have congenital abnormality
* lactose intolerant
* use antibiotic for more than 2 weeks
* consume micronutrient supplement (especially iron and zinc) in the last 3 months
* diagnose with chronic diseases and infection that interfere metabolism (i.e. tuberculosis, HIV, autoimmune disease, diabetes mellitus type 1)
* suffer marasmus and/or kwashiorkor
* not willing to continue the intervention

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-04-28 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Gut Microbiota Associated to Synbiotic Milk Treatment | 3 months
  Stools samples will be collected and analyzed before and after the intervention and compared between groups (Lactobacillus, Bifidobacteria, Bacteroides, Prevotella, and Enterobacteria) using qPCR method.

SECONDARY OUTCOMES:
Changes in Height per Age Z-score Associated to Synbiotic Milk Treatment | 3 months
  Height data will be collected and analyzed before and after the intervention and compared between groups
Changes in Hemoglobin Level Associated to Synbiotic Milk Treatment | 3 months
  Hemoglobin data will be collected and analyzed before and after the intervention and compared between groups using biochemistry method
Changes in Calprotectin Level Associated to Synbiotic Milk Treatment | 3 months
  Calprotectin data will be collected and analyzed before and after the intervention and compared between groups using immuno-assay method
Changes in Blood Zinc Level Associated to Synbiotic Milk Treatment | 3 months
  Calprotectin data will be collected and analyzed before and after the intervention and compared between groups using Atomic Absorbance Spectrophotometry method
Changes in Cognitive Level Associated to Synbiotic Milk Treatment | 3 months
  Cognitive level will be collected and analyzed before and after the intervention and compared between groups using Bayley Scales of Infant Development, 2nd Edition (BSID). This part of BSID evaluation, which yields a score called the mental development index, evaluates several types of abilities: sensory/perceptual acuities, discriminations, and response; acquisition of object constancy; memory learning and problem solving; vocalization and beginning of verbal communication; basis of abstract thinking; habituation; mental mapping; complex language; and mathematical concept formation. Total score from test will determine mental development index of children : accelerated performance (score ≥85), within normal limit (score 70-84), mildly delayed performance (score 55-69), and significantly delayed performance (score <55).
Changes in Psychomotor Level Associated to Synbiotic Milk Treatment | 3 months
  Psychomotor data will be collected and analyzed before and after the intervention and compared between groups using Bayley Scales of Infant Development, 2nd Edition (BSID). This part of the BSID assesses the degree of body control, large muscle coordination, finer manipulatory skills of the hands and fingers, dynamic movement, postural imitation, and the ability to recognize objects by sense of touch (stereognosis). Total score from test will determine motor development index of children : accelerated performance (score ≥85), within normal limit (score 70-84), mildly delayed performance (score 55-69), and significantly delayed performance (score <55).

CONTACTS AND LOCATIONS:
Overall Officials: Siti Helmyati, DR., Principal Investigator — Gadjah Mada University; Lily A. Lestari, DR., Principal Investigator — Gadjah Mada University
Locations (1):
- Universitas Gadjah Mada, Sleman, D.I.Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided